CLINICAL TRIAL: NCT00332605
Title: A Double-Blind Study of N-Acetyl Cysteine Plus Naltrexone in the Treatment of Methamphetamine Dependence
Brief Title: N-Acetyl Cysteine Plus Naltrexone in Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0601M80486
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine Dependence
MeSH Terms: interventions — Naltrexone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone plus N-Acetyl Cysteine (Experimental): Naltrexone tablets
  N-Acetyl Cysteine: 600mg tablets, daily
  Interventions: Drug: Naltrexone plus N-Acetyl Cysteine
- Placebo (Placebo Comparator): Inactive placebo ("sugar pill")
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone plus N-Acetyl Cysteine — daily
  Other Names: Naltrexone:; Revia
  Arms: Naltrexone plus N-Acetyl Cysteine
Drug: Placebo — daily
  Arms: Placebo

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of N-Acetyl Cysteine (NAC) in combination with naltrexone in methamphetamine dependence.

DETAILED DESCRIPTION:
Forty subjects with DSM-IV methamphetamine dependence will receive 8 weeks of double-blind combination medication (NAC plus naltrexone) or placebo. The hypothesis to be tested is that NAC plus naltrexone will be effective and well tolerated in patients with methamphetamine dependence compared to placebo. The proposed study will provide needed data on the treatment of a public health crisis that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 18-65
2. current DSM-IV methamphetamine dependence.

Exclusion Criteria:

1. unstable medical illness
2. history of seizures
3. myocardial infarction within 6 months
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential
5. any thoughts of suicide
6. lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder
7. previous treatment with N-Acetyl Cysteine or naltrexone
8. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline
9. abnormal liver function tests at screening
10. diagnosis of asthma
11. current use of opiates.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2006 - September 2009
Groups:
- Naltrexone: Naltrexone tablets - 50mg pills taken by mouth daily
- N-Acetyl Cysteine: 600mg tablets taken by mouth daily
- Placebo: Inactive pill taken by mouth daily
Period: Overall Study
Arm/Group | Naltrexone | N-Acetyl Cysteine | Placebo
Started | 14 | 14 | 17
Completed | 12 | 12 | 9
Not Completed | 2 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | N-Acetyl Cysteine | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 17 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 17 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (8.2) | 37.2 (8.1) | 36.1 (6.6) | 36.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 15
  Male | 8 | 8 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 17 | 45

OUTCOME MEASURES:

1. Primary Outcome: Penn Craving Scale
Description: used to measure cravings to use drugs over the past week. Range of TOTAL scores is 0-30. A lower score indicates a better outcome, while a higher score indicates a worse outcome.
Time Frame: beginning and at each visit until the end of their participation in the study
Population: Reported scores are Mean and standard deviation for Subjects last visit (including last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Naltrexone: Naltrexone tablets
- N-Acetyl Cysteine: 600mg tablets, daily
- Placebo: Placebo capsules
Arm/Group | Naltrexone | N-Acetyl Cysteine | Placebo
Number analyzed (Participants) | 14 | 14 | 17
units on a scale | 24.0 (5.5) | 24.0 (5.4) | 21.1 (6.9)

ADVERSE EVENTS:
Arm/Group | Naltrexone | N-Acetyl Cysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 8/14 | 8/14 | 7/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=14) | N-Acetyl Cysteine (N=14) | Placebo (N=17)
Nausea (Gastrointestinal disorders) | 8 (8) | 8 (8) | 7 (7)
Lethargy (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No